CLINICAL TRIAL: NCT04598022
Title: Revealing Microbiome Association With (Plant-based) Diet in Freshman
Acronym: Freshman
Status: Recruiting | Type: Observational
Sponsor: University of Kiel (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dr. Anja Bosy-Westphal, Prof. Anja Bosy-Westphal, PhD, MD, University of Kiel
Other Study IDs: ABW-2020-HM
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: freshman; vegan; vegetarian; omnivore; microbiome; meal frequency; meal timing; freshman weight gain; metabolome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum and plasma samples, saliva, urine and stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- vegan: subjects having a vegan nutrition pattern for at least the last 3 months
  Interventions: Other: cross-sectional observation; Other: cross-sectional follow-up observation
- vegetarian: subjects having a vegetarian nutrition pattern for at least the last 3 months
  Interventions: Other: cross-sectional observation; Other: cross-sectional follow-up observation
- omnivores: subjects having a omnivore nutrition pattern for at least the last 3 months
  Interventions: Other: cross-sectional observation; Other: cross-sectional follow-up observation

INTERVENTIONS:
Other: cross-sectional observation — observation of dietary patterns, body weight status, microbiome and metabolome profiles at the start of the first semester
Other: cross-sectional follow-up observation — follow-up observation of dietary patterns, body weight status,microbiome and metabolome profiles after one year

SUMMARY:
Aim of the study is to evaluate the impact of a vegan vs. vegetarian dietary pattern compared to an omnivore diet on body weight, saliva and stool microbiome profiles, as well as saliva, urine and plasma metabolome profile changes in freshmen after the first year at university/college.

ELIGIBILITY:
Inclusion Criteria:

* freshman
* following a vegan / vegetarian / omnivore dietary pattern for at least 3 months
* own a smartphone (including internet access and camera)

Exclusion Criteria:

* regular use of medication (excluding oral contraceptiva)
* use of antibiotics in the last 6 weeks
* chronic disease, especially gut diseases
* following a vegan / vegetarian / omnivore dietary pattern for less then 3 months
* no clear assignment of vegan / vegetarian / omnivore dietary pattern
* electrical implants

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy university / college freshmen studying in Kiel, Germany
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
change in body weight | one year
  change in body weight
change in fat mass | one year
  change in body composition

SECONDARY OUTCOMES:
saliva metabolome | one year
  changes in saliva metabolome
gut microbiome | one year
  changes in gut microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Anja Bosy-Westphal, PhD, MD, Principal Investigator — Institute of Human Nutrition, Kiel University
Locations (1):
- Institute of Human Nutrition, Kiel, Germany